CLINICAL TRIAL: NCT00902382
Title: Registry of Pregnancies Conceived Following Exposure to Ovulation Stimulation Medications
Status: Completed | Type: Observational
Sponsor: Yale University (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH); Penn State University (Other); University of Colorado, Denver (Other); University of Michigan (Other); University of Pennsylvania (Other); University of Texas (Other); University of Vermont (Other); Wayne State University (Other)
Responsible Party: Principal Investigator, Heping Zhang, Principal Investigator, Yale University
Other Study IDs: RMN-PregReg; RMN Pregnancy Registry
Record Dates: First submitted 2009-05-13; First posted 2009-05-15 (Estimated); Last update posted 2018-02-07 (Actual); Status verified 2018-02

CONDITIONS: Infertility
Keywords: Infertility; Ovulation stimulation; Pregnancy
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Mothers of newborn infants will be asked to consent to the collection of buccal cells from their infants for DNA testing. Fathers will also be asked to provide buccal cells via buccal swab smears, if blood has not been obtained from them in the course of an RMN trial. The DNA specimens will be available for use in other vetted studies to enable study of independent genetic and environmental factors and gene-environment interactions for a broad range of birth defects and infertility.
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- 1: Infertile women who conceive spontaneously
- 2: Infertile women who conceive on various ovulation stimulation medications

SUMMARY:
To identify adverse effects of ovulation drugs on pregnancy, including pregnancy loss, fetal teratology and dysmorphology, and infant development up to age 3.

DETAILED DESCRIPTION:
This will be an observational cohort trial of the pregnancy of women who conceive in RMN trials, and of their resulting infants through the first 3 years of life.

Study specific procedures will include a patient completed log of prescribed and over the counter medications taken during a normal pregnancy, a review of their pregnancy, delivery, and neonatal records, an exam of the infant within 60 days of birth by a dysmorphologist, and yearly review of infant medical records, growth charts, and a yearly parent administered developmental questionnaire (Ages and Stages) for the first three years of the infant's life.

ELIGIBILITY:
Inclusion Criteria:

* Positive serum hCG within the context of a RMN trial;
* History of infertility meeting female subject entry criteria for a RMN trial;
* Informed consent.

Exclusion Criteria:

* Unable to comply with the demands of the trial.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: The population will include women with infertility who receive ovulation stimulation drugs within the context of a Reproductive Medicine Network sponsored trial as well as their infants.
Sampling Method: Non-Probability Sample
Enrollment: 264 (Actual)
Dates: Start 2009-05; Primary Completion 2014-06-27 (Actual); Study Completion 2014-06-27 (Actual)

PRIMARY OUTCOMES:
The relative risks of genetic abnormalities identified at birth and within the first 60 days of life | 2009 - 2016
The relative risk of structural anomalies | 2009 - 2016
The relative risk of cognitive differences | 2009 - 2016
The relative risk of perceived differences of neuro-developmental milestones | 2009 - 2016

SECONDARY OUTCOMES:
The rate of pregnancy complications, including pregnancy loss | 2009 - 2016
Rates of neonatal and infant medical disorders | 2009 - 2016
Rates of infant growth related to use of letrozole for stimulation of ovulation compared to other treatment modalities for ovulation stimulation, including compared to women who conceive spontaneously. | 2009 - 2016

CONTACTS AND LOCATIONS:
Overall Officials: Esther Eisenberg, MD, MPH, Principal Investigator — Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD); Nanette Santoro, MD, Study Chair — Albert Einstein College of Medicine; Richard Legro, MD, Principal Investigator — Pennsylvania State University College of Medicine; Robert Brzyski, MD, PhD, Study Director — The University of Texas Health Science Center at San Antonio; Peter Casson, MD, Study Director — University of Vermont; Michael Diamond, MD, Principal Investigator — Wayne State University; Heping Zhang, PhD, Study Director — Yale University; Gregory Christman, MD, Study Director — University of Michigan; Christos Coutifaris, MD, Study Director — University of Pennsylvania; William Schlaff, MD, Study Director — University of Colorado Denver Health Science Center
Locations (13):
- United States (13):
  - University of Alabama Birmingham, Birmingham, Alabama
  - Stanford University Medical Center, Stanford, California
  - University of Colorado, Aurora, Colorado
  - Yale University, New Haven, Connecticut
  - University of Michigan, Ann Arbor, Michigan
  - Wayne State University, Detroit, Michigan
  - Hackensack University, Hackensack, New Jersey
  - Carolinas Medical Center, Charlotte, North Carolina
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Pennsylvania State University College of Medicine, Hershey, Pennsylvania
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas
  - University of Vermont, Burlington, Vermont